CLINICAL TRIAL: NCT04416594
Title: Impact of Acquired FXIII Deficiency on Morbidity and Mortality Among Hospitalized Patients
Brief Title: Impact of Acquired FXIII Deficiency on Morbidity and Mortality
Status: Completed | Type: Observational
Sponsor: Patricia Duque González (Other)
Responsible Party: Sponsor-Investigator, Patricia Duque González, Principal Investigator, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Other Study IDs: FXIII
Record Dates: First submitted 2020-05-26; First posted 2020-06-04 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Acquired Factor XIII Deficiency Disease
Keywords: Factor XIII; Blood transfusion; Mortality
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Factor XIII deficiency: Patients admitted to hospital with FXIII levels below 70% during their hospital stay
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Only data collection

SUMMARY:
Observational prospective study aiming to assess acquired FXIII deficiency implications in morbidity and mortality

DETAILED DESCRIPTION:
All patients admitted to a large tertiary hospital with FXIII levels below 70% during their hospital stay are assessed. Data regarding patient background, blood transfusion, morbidity and mortality is registered.

ELIGIBILITY:
Inclusion Criteria:

* FXIII levels < 70%

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Medical and surgical hospitalized patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
Cut-Point levels of FXIII | 2 years
  The investigators aim to find a laboratory parameter, a cut-point plasma level of FXIII, to identify an increased in morbidity and mortality in a mixed cohort of hospitalized patients

CONTACTS AND LOCATIONS:
Locations (1):
- Gregorio Marañon Hospital, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Duque P, Esteban ML, Pineiro P, Ortiz-Lopez A, Moreno-Carbonell M, Lancho P, Calvo A, Terradillos E, Pascual-Izquierdo C. Acquired factor XIII deficiency is associated with mortality and is not linked to hypocalcemia. Blood Coagul Fibrinolysis. 2026 Jan 1;37(1):28-37. doi: 10.1097/MBC.0000000000001400. Epub 2025 Nov 27. PMID 41311329
- [Derived] Duque P, Chasco-Ganuza M, Ortuzar A, Almaraz C, Terradillos E, Perez-Rus G, Pascual C. Acquired FXIII Deficiency is Associated with High Morbidity. Thromb Haemost. 2022 Jan;122(1):48-56. doi: 10.1055/a-1481-2733. Epub 2021 Jun 6. PMID 33851388